CLINICAL TRIAL: NCT01340183
Title: A Phase I, Single-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics in Intravenous AZD5099 After Single Ascending Doses in Healthy Male and Female Subjects
Brief Title: Clinical Study Assessing the Safety, Tolerability, and Pharmacokinetics of Intravenous AZD5099 in Healthy Subjects
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: D0910C00015
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Phase I; safety; tolerability; pharmacokinetics; AZD5099; volunteers; safety of the drug AZD5099; blood and urine levels of AZD5099; single intravenous doses; healthy volunteers
MeSH Terms: interventions — 2-(4-((3,4-dichloro-5-methyl-1H-pyrrole-2-carbonyl)amino)-3-methoxy-1-piperidyl)-4-((2-methoxy-1-methylethyl)carbamoyl)thiazole-5-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AZD5099 (Experimental): IV Dose
  Interventions: Drug: AZD5099
- Placebo (Placebo Comparator): IV Dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5099 — IV Dose
  Arms: AZD5099
Drug: Placebo — IV Dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of the drug AZD5099 after intravenous administration of single doses in healthy volunteers. The results from this study will form the basis for decisions regarding the future development of AZD5099 as a novel antibiotic for the treatment of serious infections in humans.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures including the genetic sampling
* Healthy male and female (with nonchildbearing potential) volunteers aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of nonchildbearing potential, confirmed at screening by fulfilling 1 of the following criteria:
* Postmenopausal, defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with follicle stimulating hormone (FSH) levels within the laboratory-defined post-menopausal range
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation
* Male volunteers should be willing to use barrier contraception, ie, condoms, from the day of dosing until at least 3 months after dosing with the investigational product
* Have a body mass index (BMI) between 18 and 30.5 kg/m2 and weigh at least 50 kg and no more than 100 kg inclusive

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product
* History of gastrointestinal ulcer disease, inflammatory bowel disease, indigestion symptoms >3 times a week, or blood in stool in previous 6 months not related to anal trauma
* For male volunteers any history of sexual dysfunction or impotence as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD5099 | Ongoing throughout the study from consent (up to 28 days prior to dosing) through withdrawal or completion (up to 10 days after discharge).
  To assess the safety and tolerability of AZD5099 by documenting: 1) the incidence and severity of adverse events, 2) abnormalities and time matched comparison from Day -1 to Day 1 of core body temperature and vital sign assessments, 3) electrocardiograms (ECGs), 4) telemetry, 5) clinical laboratory assessments, 6) physical examinations, and 7) withdrawals.

SECONDARY OUTCOMES:
Blood samples to characterize the pharmacokinetics of AZD5099, pre-dose | Pre-dose
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 15 min | 15 minutes post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 30 min | 30 minutes post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 1 hour | 1 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 2 hour | 2 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 2.5 hour | 2.5 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 3 hour | 3 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 4 hour | 4 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 5 hour | 5 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 6 hour | 6 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 8 hour | 8 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 10 hour | 10 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 12 hour | 12 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 24 hour | 24 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 36 hour | 36 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 48 hour | 48 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 72 hour | 72 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 96 hour | 96 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Blood samples to characterize the pharmacokinetics of AZD5099, 120 hour | 120 hour post start of infusion
  Blood samples will be taken to characterize the pharmacokinetics of AZD5099 by determination of Cmax, tmax, λz, AUC, AUC(0-t), t½λz, Vz, Vdss, and CL.
Urine samples to characterize the pharmacokinetics of AZD5099, pre-dose | Between -12 to 0 hours
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 0-4 hours | Between 0 - 4 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 4-8 hours | Between 4 - 8 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 8-12 hours | Between 8 - 12 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 12-24 hours | Between 12 - 24 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 24-48 hours | Between 24 - 48 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 48-72 hours | Between 48 - 72 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 72-96 hours | Between 72 - 96 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].
Urine samples to characterize the pharmacokinetics of AZD5099, 96-120 hours | Between 96 - 120 hours post start of infusion
  Urine samples to characterize the pharmacokinetics of AZD5099 by determination of the cumulative amount of unchanged drug excreted in urine [Ae(0-t)], and fraction of dose excreted into urine [fe(0-t)].

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, MD, Principal Investigator — Parexel; David Melnick, Study Director — AstraZeneca
Locations (1):
- Research Site, Glendale, California, United States